CLINICAL TRIAL: NCT02404454
Title: Prevention of Intrauterine Adhesions After Hysteroscopic Metroplasty With Autocross-linked Hyaluronic Acid Gel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Università degli Studi di Sassari (Other); Azienda Sanitaria Locale di Cagliari (Other); Azienda Sanitaria Locale di Olbia (Other); Azienda Sanitaria Locale di Oristano (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MulticentricMetroplasty
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Intrauterine Adhesions; Septate Uterus
MeSH Terms: conditions — Gynatresia; Septate Uterus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hysteroscopic metroplasty (Experimental): women undergoing hysteroscopic metroplasty for uterine septum resection
  Interventions: Procedure: Hysteroscopic metroplasty; Device: Autocross-linked acid hyaluronic gel; Procedure: Office second look hysteroscopy

INTERVENTIONS:
Procedure: Hysteroscopic metroplasty
Device: Autocross-linked acid hyaluronic gel — Patients received adhesion barrier with 5 ml of autocross-linked acid hyaluronic gel
Procedure: Office second look hysteroscopy — Second-look hysteroscopy after three months

SUMMARY:
The septate uterus is the most common structural uterine anomaly. It results from failure of the partition between the two fused Müllerian ducts to resorb;it is associated with the highest incidence of reproductive failure and with first- and second-trimester pregnancy loss and infertility.

Hysteroscopic division of the uterine septum is performed using microscissors, electrosurgery, or laser. Several studies shown significant improvement in pregnancy outcome after hysteroscopic metroplasty.

Purpose of this study is to verify the effectiveness of 5 ml, instead of 10 ml, of autocross-linked hyaluronic acid gel in the prevention of the formation of intrauterine adhesions, through second look office hysteroscopy after three months.

ELIGIBILITY:
Inclusion Criteria:

* uterine septum
* history of ≥1 miscarriage or infertility;
* desire to have children in the future

Exclusion Criteria:

* pregnancy;
* menopause;
* precancerous state or malignancy of the reproductive organs;
* benign lesions in the myometrium of the uterine fundus (myomas or adenomyosis)
* lesions distorting the uterine cavity (submucosal myomas or intrauterine adhesions) on ultrasonography;
* withdrawal of patient consent;
* rare complex uterine congenital anomalies without an ASRM classification such as uterine septum with double cervix ;
* presence of external intercornual cleft;
* incomplete (internal fundal indentation 10 mm) or non-standardized septum resection (internal fundal indentation ,10 mm and uterine myometrial thickness .10 mm at the fundus), confirmed intraoperatively
* excessive fundal incision (uterine myometrial thickness ,6 mm at the fundus confirmed intraoperatively)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in Formation of intrauterine adhesions | baseline (operative isteroscopy and three months